CLINICAL TRIAL: NCT00886613
Title: A Double-Blind, Randomized, Placebo Controlled, Parallel Group Study to Evaluate Biomarkers of Immunity to Varicella Zoster Virus Following Immunization With V212/Heat-Treated Varicella-Zoster Virus (VZV) Vaccine or With ZOSTAVAX in Healthy Volunteers
Brief Title: A Study to Evaluate Immunity to Varicella Zoster Virus After Immunization With V212 Vaccine or Zostavax (V212-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V212-003; 2009_579
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2011-04-13 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- V212 (Experimental): Participants randomized to receive V212 (heat treated VZV Vaccine)
  Interventions: Biological: V212; Other: VZV Skin Test; Other: Saline
- Zostavax™ (Active Comparator): Participants randomized to receive Zostavax™ (Zoster Vaccine, live)
  Interventions: Biological: Comparator: Zostavax™; Other: VZV Skin Test; Other: Saline
- Placebo (Placebo Comparator): Participants randomized to receive placebo
  Interventions: Biological: Comparator: Placebo; Other: VZV Skin Test; Other: Saline

INTERVENTIONS:
Biological: V212 — Two doses of 0.65 mL V212 subcutaneous injection administered at Day 1 and Day 31
  Arms: V212
Biological: Comparator: Zostavax™ — Two doses of 0.65 mL Zostavax™ subcutaneous injection administered at Day 1 and Day 31
  Other Names: V211 (Zoster Vaccine Live (Oka/Merck))
  Arms: Zostavax™
Biological: Comparator: Placebo — Two doses of 0.65 mL subcutaneous injection of placebo administered at Day 1 and Day 31
  Arms: Placebo
Other: VZV Skin Test — Three intradermal injections of the 0.1 ml varicella antigen (VZV Skin Test reagent) were administered, once at baseline before the first vaccination, a second time before the second vaccination, and a third time approximately 14 days after the second vaccination.
Other: Saline — One intradermal injection of the 0.1 ml saline was administered at the time of the baseline VZV skin test prior to the first vaccination. Saline and VZV skin test reagents were administered on opposite arms.

SUMMARY:
A study in two parts (Part A and Part B) to evaluate the responsiveness of various biomarkers of immunity to Varicella-Zoster Virus (VZV) following repeated immunizations with heat treated VZV vaccine V212 or with Zostavax™.

The enrollment of participants into this study was conducted in 2 parts, Part A and Part B. The first 42 eligible participants were enrolled into Part A of the study. In Part A, the reaction of the VZV skin test at baseline was evaluated at both 48 and 72 hours post administration of the VZV skin test reagent and saline (in opposite arms), with 2 examiners performing the reading at each timepoint; all subsequent skin test readings in Part A were performed at 48 hours post administration. After all skin test reactions were obtained at baseline for the 42 subjects in Part A, an interim analysis was performed (1) to assess the frequency of baseline negative skin tests in order to confirm that the planned sample size (N=120) was adequate for an evaluation of the effect of vaccination on the VZV Skin Test, and (2) to assess the frequency of baseline positive skin tests at 72 hours relative to 48 hours (post administration) in order to determine the preferred time for evaluation of the skin test reaction.

The interim analysis from Part A confirmed the study sample size, an additional 78 subjects were enrolled into Part B to achieve the planned sample size (N=120). The study procedures for Part B of the study were identical to those in Part A with the following exceptions: (1) baseline skin test readings were performed only once, at either 48 or 72 hours (post administration) to accommodate the scheduling of clinic visits, and (2) only one examiner was needed for the skin test reading at baseline.

DETAILED DESCRIPTION:
All eligible participants, regardless of treatment group, were administered three injections of the varicella antigen (VZV Skin Test reagent), once at baseline before the first vaccination, a second time before the second vaccination, and a third time approximately 14 days after the second vaccination. Reactions to the skin test were assessed by the same examiner for each participant to the greatest extent possible.

ELIGIBILITY:
Inclusion Criteria:

* Participant has prior history of Varicella
* Female participants are of non-childbearing potential

Exclusion Criteria:

* Participant has had a hypersensitivity reaction to any vaccine component
* Participant has a prior history of Herpes Zoster
* Participant has received any Varicella or Zoster vaccine including Zostavax
* Participant has a history of immunosuppression caused by disease, corticosteroids, cancer therapy or organ transplant
* Participant has an active cancer
* Participant has received or will receive a live virus vaccine or an inactivated virus vaccine 4 weeks prior to participating in study (with the exception of influenza vaccine)
* Participant is not bed-ridden or homebound

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed in 2 parts - Part A and Part B, with a total of 120 participants.
Pre-assignment Details: In Part A, 42 participants received a baseline VZV Skin Test which was evaluated 48 and 72 post administration, and these participants were included in the analysis for Part B. All Participants were randomized to receive V212, Zostavax™ or placebo.
Groups:
- V212: Participants randomized to receive two subcutaneous injections of 0.65 mL V212 (heat treated VZV Vaccine)
  administered at Day 1 and Day 31.
- Zostavax™: Participants randomized to receive two subcutaneous injections of 0.65 mL Zostavax™ administered at Day 1 and Day 31.
- Placebo: Participants randomized to receive two subcutaneous injections of 0.65 mL of placebo administered at Day 1 and Day 31.
Period: Overall Study
Arm/Group | V212 | Zostavax™ | Placebo
Started | 41 | 39 | 40
Completed | 39 | 39 | 37
Not Completed | 2 | 0 | 3
Not completed — Protocol deviation (Part B) | 1 | 0 | 0
Not completed — Lost to follow-up (Part B) | 1 | 0 | 1
Not completed — Subject withdrew consent (Part A) | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V212 | Zostavax™ | Placebo | Total
Number analyzed (Participants) | 41 | 39 | 40 | 120
Age, Customized [Number; unit: participants]
  Between 60 and 88 years | 41 | 39 | 40 | 120
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 23 | 74
  Male | 16 | 13 | 17 | 46
Region of Enrollment [Number; unit: participants]
  United States | 41 | 39 | 40 | 120

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Number of Participants With a Negative Reaction for Saline at Baseline (Part A)
Description: Participants were given the VZV skin test prior to vaccination. For the baseline VZV skin test, they were administered VZV skin test reagent and saline in opposite arms. The skin reaction (erythema and induration) to saline was marked with a ball point pen. The longest dimension to the closest 1 mm was measured. Participants with a reaction measure < 5mm for saline had a negative reaction for saline, and measure >= 5mm for saline had a positive reaction for saline at baseline.
Time Frame: 48 hours following administration of the baseline skin test
Population: 42 participants enrolled in Part A
Measure: Number; unit: Participants
Groups:
- Part A Participants - VZV Skin Reaction (Baseline): All 42 participants enrolled for part A were administered the VZV skin test and assessed for a skin reaction at baseline.
Arm/Group | Part A Participants - VZV Skin Reaction (Baseline)
Number analyzed (Participants) | 42
Participants
  Negative reaction to saline | 39
  Positive reaction to saline | 2
  Participants with missing assessment | 1

2. Primary Outcome: Number of Participants With a Negative VZV Skin Test at Baseline (Part A)
Description: Participants were given the VZV skin test prior to vaccination. For the baseline VZV skin test, they were administered VZV skin test reagent and saline in opposite arms, and assessed for a skin reaction around the injection site. The skin reaction assessed was erythema (redness of skin) and induration (palpable, raised, hardened area) around the injection site, which was marked with a ball point pen. The longest dimension to the closest 1 mm was measured. Participants with a reaction measure < 5mm for saline and < 5mm for the VZV antigen were considered to have a negative baseline skin test.
Time Frame: 48 hours following administration of the baseline skin test
Population: Participants enrolled in Part A with a negative reaction for saline.
Measure: Number; unit: Participants
Arm/Group | Part A Participants - VZV Skin Reaction (Baseline)
Number analyzed (Participants) | 39
Participants | 23

3. Secondary Outcome: VZV Skin Test Reactions at 48 and 72 Hours (Part A)
Description: Prior to vaccination, participants were administered a baseline VZV skin test for which the skin test reagent and saline were injected in opposite arms. The skin reaction (erythema and induration) around the injection site was assessed at 48 hours and at 72 hours. The reaction was marked with a ball point pen and the longest dimension closest to 1 mm was measured. Participants with a reaction measure < 5mm for saline and < 5mm for the VZV antigen were defined as having a negative baseline skin test; and a measure of >= 5mm for the VZV antigen were defined as having a positive skin test.
Time Frame: 48 hours and 72 hours post administration of baseline skin test
Population: 42 participants enrolled in Part A
Measure: Number; unit: Participants
Groups:
- Part A Participants - VZV Skin Reaction (48 Hrs): All 42 participants enrolled for part A were administered the VZV skin test and assessed for a skin reaction after 48 hours.
- Part A Participants - VZV Skin Reaction (72 Hrs): All 42 participants enrolled for part A were administered the VZV skin test and assessed for a skin reaction after 72 hours.
Arm/Group | Part A Participants - VZV Skin Reaction (48 Hrs) | Part A Participants - VZV Skin Reaction (72 Hrs)
Number analyzed (Participants) | 42 | 42
Participants
  Participants with a negative VZV skin test | 24 | 25
  Participants with a positive VZV skin test | 18 | 17
Statistical Analysis 1: Comparison: Part A Participants - VZV Skin Reaction (48 Hrs) vs Part A Participants - VZV Skin Reaction (72 Hrs); Test type: Superiority or Other; p = 0.564, McNemar; kappa coefficient of agreement = 0.85, 90% CI 2-sided [0.72 to 0.99] — The significance of the difference between the proportion of subjects with a positive skin test at 48 hours and the proportion of subjects with a positive skin test at 72 hours

4. Secondary Outcome: Number of Healthy Elderly Men and Women With Adverse Events Post Vaccination With V212 (Part B)
Description: The number of participants with all serious and nonserious adverse events, and vaccine-related serious and nonserious adverse events, from 1-28 days post any vaccination dose was determined to assess safety. Non serious adverse events include injection-site adverse events as well as systemic adverse events post vaccination. Vaccine-related events include all events that were possibly, probably or definitely related to the vaccine according to the investigator. Participants with injection site adverse events due to administration of VZV skin tests are not included.
Time Frame: 1-28 days post vaccination dose 1 and 1-28 days post vaccination dose 2
Population: Participants from Part B. One participant in the placebo group was not vaccinated and is not included in the analysis.
Measure: Number; unit: Participants
Arm/Group | V212 | Zostavax™ | Placebo
Number analyzed (Participants) | 41 | 39 | 39
Participants
  No adverse experiences (AE) | 17 | 10 | 10
  One or more AE | 22 | 26 | 19
  One or more injection-site AE | 11 | 26 | 9
  One or more systemic AE | 15 | 14 | 14
  One or more vaccine-related (VR) AE | 12 | 24 | 9
  One or more VR injection-site AE | 11 | 22 | 8
  One or more VR systemic AE | 1 | 5 | 2
  One or more SAE | 0 | 0 | 0
  One or more VR SAE | 0 | 0 | 0

5. Primary Outcome: Number of Healthy, Elderly, Immunocompetent Participants With a Positive VZV Skin Test After Administration of 2 Doses of V212 Vaccine (Part B)
Description: Number of participants with a positive VZV skin test after 2 vaccine doses was determined. Participants with a negative VZV skin test reaction at baseline were evaluated for VZV immunogenicity by a final VZV skin test administered 14 days after dose 2 of vaccination.
  For the VZV skin test participants were injected intradermally with the VZV skin test reagent, and reaction to the skin test was assessed after 48-72 hrs. A skin reaction (erythema and induration) around the injection site measuring >= 5mm for the VZV antigen was considered a positive skin test.
Time Frame: 48-72 hours after administration of skin test at 14-17 days postdose 2
Population: Per protocol population - participants with a negative baseline VZV Skin Test (<5 mm skin reaction to both, saline and the VZV skin test reagent), and who did not have a protocol deviation that could interfere with the immune response to vaccine following two administrations of either ZOSTAVAX™, placebo, or V212
Measure: Number; unit: Participants
Arm/Group | V212 | Zostavax™ | Placebo
Number analyzed (Participants) | 28 | 28 | 25
Participants | 15 | 15 | 12
Statistical Analysis 1: Comparison: V212 vs Placebo; Test type: Superiority or Other; p = 0.343, Chi-squared; Difference in proportions = 0.06, 90% CI 2-sided [-0.17 to 0.28] — Statistical analysis for dose 2

6. Secondary Outcome: Number of Healthy Elderly Men and Women With Injection Site Adverse Events Post Administration of VZV Skin Tests (Part B)
Description: The number of participants with injection site adverse events due to the VZV skin test after administration of the VZV skin test antigen.
Time Frame: 1-5 days post administration of each VZV skin test
Population: Participants from Part B. One participant in the placebo group was not vaccinated and is not included in the analysis.
Measure: Number; unit: Participants
Arm/Group | V212 | Zostavax™ | Placebo
Number analyzed (Participants) | 41 | 39 | 39
Participants | 36 | 36 | 28

ADVERSE EVENTS:
Time Frame: 1-28 days post any vaccine dose
Description: The analyzed population includes all vaccinated participants. One participant in the placebo group was not vaccinated and is not included in the analysis.
Arm/Group | V212 | Zostavax™ | Placebo
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 36/41 | 36/39 | 29/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | V212 (N=41) | Zostavax™ (N=39) | Placebo (N=39)
Headache (Nervous system disorders) | 1 | 2 | 2
Injection site erythema (Vaccination) (General disorders) | 11 | 18 | 7 — Injection site reaction following administration of V212, Zostavax™ or placebo.
Injection site erythema (Skin test) (General disorders) | 36 | 36 | 28 — Injection site reaction following administration of the skin test.
Injection site induration (Vaccination) (General disorders) | 6 | 16 | 4 — Injection site reaction following administration of V212, Zostavax™ or placebo.
Injection site induration (Skin test) (General disorders) | 19 | 18 | 17 — Injection site reaction following administration of the skin test.
Injection site pain (Vaccination) (General disorders) | 4 | 21 | 2 — Injection site reaction following administration of V212, Zostavax™ or placebo.
Injection site pain (Skin test) (General disorders) | 5 | 8 | 2 — Injection site reaction following administration of the skin test.
Injection site pruritis (Vaccination) (General disorders) | 2 | 2 | 0 — Injection site reaction following administration of V212, Zostavax™ or placebo.
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multicenter studies, an investigator and his/her colleagues may publish their data independently subsequent to the multicenter publication. The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. SPONSOR review can be expedited to meet publication timelines.